CLINICAL TRIAL: NCT05736666
Title: Preoperative Perturbation Training to Prevent Falls After Total Knee Arthroplasty
Brief Title: Treadmill Perturbation Training for Fall Prevention After Total Knee Replacement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kharma C Foucher, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-0366; R01AG075098 (NIH)
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Knee Osteoarthritis; Arthroplasty Complications
Keywords: Falls; Knee Replacement
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): The intervention consists of disturbances delivered on a treadmill that simulates tripping over an obstacle or being perturbed to the side.
  Interventions: Behavioral: Treadmill-based perturbation training
- Education Group (Active Comparator): This group will receive educational materials related to fall prevention in older adults.
  Interventions: Behavioral: Education Control

INTERVENTIONS:
Behavioral: Treadmill-based perturbation training — The intervention consists of disturbances delivered on a treadmill that simulates tripping over an obstacle or being perturbed to the side. These disturbances require a compensatory step to respond. Through this task-specific training, participants should learn to control their trunk motion in a way that will cause them to avoid a trip or fall to the side.
  Arms: Training Group
Behavioral: Education Control — Fall prevention educational material
  Arms: Education Group

SUMMARY:
The goal of this clinical trial is to learn about preventing falls in people who have total knee replacement surgery using treadmill perturbation training. Perturbation training involves adjusting to rapid speed changes on a treadmill. The main questions it aims to answer are:

* Does perturbation training improve the way that people who are planning to have total knee replacement surgery recover after treadmill test that reproduces a trip to the front or side?
* Does perturbation training reduce the incidence of preventable gait-related falls during the first year after total knee replacement?

Participants will:

* complete surveys about their condition and fall history and take part in testing of walking ability and balance.
* have a baseline gait analysis test to measure the motion of their body during normal walking.
* Be randomized into two groups. One will receive fall-prevention literature. The other will receive the same literature and then take part in a two-week treadmill perturbation training program.
* be contacted every two weeks for one year, and asked questions about whether they have fallen during that time.
* wear a Fitbit activity monitor on their wrist for one year. Researchers will compare the number of falls from the group that only received literature to the treatment group to see if the training group has fewer falls during the year after surgery.

DETAILED DESCRIPTION:
Participants:

We will recruit 196 participants who are scheduled for primary unilateral total knee arthroplasty (TKA) and can commit to 5 additional study visits.

Baseline assessment: At enrollment, all participants will be assessed for a set of demographic and functional risk factors listed below

1. Age
2. Sex
3. Body mass index
4. Number of painful joints - Patient Reported Arthralgia Inventory
5. Medications that increase fall risk
6. Number of falls in the past 12 months
7. Self-reported activity level (UCLA activity score)
8. Habitual walking speed (8-meter walk test)
9. Functional Limitations

   1. PROMIS (Patient-Reported Outcomes Measurement Information Systems) Physical Function computerized adaptive test (CAT)
   2. Knee Injury and Osteoarthritis Outcome Score (KOOS) Activities of Daily Living Subscale
10. Pain - KOOS pain subscale; Intermittent and Constant Osteoarthritis Pain Scale; Pain Catastrophizing Scale; Tampa Scale of Kinesiophobia
11. Balance and mobility impairment

    1. Timed up and go test
    2. 30 second chair stand test
    3. 4 stage balance test
    4. 8 m walk test
    5. Functional reach test
    6. 6-minute walk test
    7. 4 square step test
12. Comorbidities - SCQ comorbidity questionnaire
13. Depression - PROMIS depression (CAT)

Participants will also undergo a standard gait analysis assessment consisting of approximately 5 nonconsecutive minutes of walking at comfortable and fast speeds on an instrumented treadmill with reflective markers will be placed on bony landmarks of the trunk, arms, and lower extremities.

After this assessment, participants will be provided with a Fitbit that they will wear daily except during bathing or swimming. Physical activity level will be measured for the duration of the follow-up period (1 year).

Finally, randomization assignments will be provided along with written education materials (fall prevention brochures from the Centers for Disease Control and Prevention), and the following activities will be undertaken according to grouping:

Group 1 - Perturbation training (4 sessions over 2 weeks with a post-test session 1 week later):

1. 30 reflective markers will be placed on bony landmarks of the trunk, arms, and lower extremities with one marker indicating the proximal and distal end of each segment and one marker placed out of line with the other two so that the motion capture software can define the 3D motion of each segment.
2. Participants will be stand comfortably with feet at approximately hip width, on a split belt treadmill. They will be fitted with a safety harness. They will be instructed that the treadmill will move and that they should do whatever they can to maintain or regain their balance.
3. During the next one minute, a tester will activate the treadmill. Two small surface translations (0.02 cm at roughly 0.22 m/s) will then be administered which will require several small forward directed steps to regain stability. These two small disturbances will provide a familiarization of how the treadmill works.
4. Participants will be informed that they will receive up to 30 disturbances of larger magnitude while facing forward, then again while facing to each side. They will be instructed to "do whatever [they] can to recovery [their] balance".
5. On the next perturbation, the participant will receive a larger disturbance. Each training perturbation will consist of the treadmill accelerating for 300 ms, maintaining a constant velocity for 170 ms, then decelerating to 0 m/s in 100 ms. Prior to the disturbance participants will be informed to recover their balance and continue walking for 5 seconds after the perturbation.
6. The tester will then administer no more than 30 disturbances of increasing difficulty as tolerated by the participant.
7. A final perturbation will be administered. This constitutes the post-test assessment.
8. Steps 2-7 will be repeated with the participant turned 90 degrees such that a step to the side will be required. The magnitude of the perturbations will be scaled to 2 foot widths.
9. Step 8 will be repeated with the participant turned by 180 degrees such that both sides receive lateral training.

Group 2 - Education Control: this group will not undergo additional training but will only receive the written materials

Beginning one week after surgery and then every two weeks for one year, participants will be contacted by text message and asked whether they had fallen during the previous two weeks. People who report falls will be contacted for a detailed interview about the circumstances and consequences of the event.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of endstage knee osteoarthritis requiring total knee arthroplasty (TKA). TKA scheduled within two months and able to schedule the required training visits prior to surgery.

Exclusion Criteria: Potential participants will be excluded if they have dizziness or self-reported medical conditions that would be expected to affect walking and balance. These specifically include history of stroke, multiple sclerosis, Parkinson's disease, and balance disorders including positional vertigo and Meniere's disease. Other exclusion criteria include plans to undergo a contralateral TKA within 12 months or history of other lower extremity joint replacement within 5 years. Finally, people who report idiopathic low back pain, history of heart disease, uncorrected vision impairment, or institutionalization will be excluded.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Post-training trunk angle | Immediately after completion of training program
  post-training trunk angle at recovery step completion
Post-training trunk angular velocity | Immediately after completion of training program
  post-training trunk angular at recovery step completion
Fall rate | 1 year
  Number of falls during the first year after surgery

SECONDARY OUTCOMES:
Fall status | Immediately after completion of training program
  Did participant fall during the post-training test

CONTACTS AND LOCATIONS:
Overall Officials: Kharma Foucher, MD, PhD, Principal Investigator — University of Illinois Chicago
Locations (1):
- Biomechanics and Clinical Outcomes Laboratory, University of Illinois Chicago, Chicago, Illinois, United States